CLINICAL TRIAL: NCT07246642
Title: Randomized Controlled Trial of Intracorporal Local Anesthesia vs Saline Prior to Placement of Inflatable Penile Prosthesis Placement
Brief Title: IPP Placement & Intracavernosal Block
Acronym: IPP
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00129597
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-09

CONDITIONS: Erectile Dysfunction (ED)
Keywords: inflatable penile prosthesis (IPP); Pain management; Penile pain
MeSH Terms: conditions — Erectile Dysfunction; Agnosia

STUDY DESIGN:
Intervention Model Description: Patients will be randomized at the time of surgery into one of two groupings: 1-10cc saline injection into each corpora for a total of 20cc immediately prior to placement of corporotomy stay sutures or 2- a 10cc of Exparel (133 mg, 1.3%) with 10cc of 0.5% standard bupivacaine (50 mg) for total volume of 20cc into the corpora immediately prior to placement of corporotomy stay sutures.
Who Masked: Participant, Care Provider
Masking Description: double blinding - the patients and the interviewing individuals
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Saline Arm (No Intervention): 10cc of normal saline will be injected into each corporal body (left and right for a total of 20cc)
- Exparel/bupivacaine mixture Arm (Experimental): 10cc Exparel/bupivacaine mixture will be injected into each corporal body (left and right for a total of 20cc)
  Interventions: Drug: Exparel/bupivacaine mixture

INTERVENTIONS:
Drug: Exparel/bupivacaine mixture — 10cc of Exparel (133 mg, 1.3%) with 10cc of 0.5% standard bupivacaine (50 mg )for total volume of 20cc into the corpora immediately prior to placement of corporotomy stay sutures.
  Other Names: Exparel (133 mg, 1.3%) with 10cc of 0.5% standard bupivacaine (50 mg)
  Arms: Exparel/bupivacaine mixture Arm

SUMMARY:
The inflatable penile prosthesis (IPP) is the gold standard for surgical management of erectile dysfunction (ED) and there is no consensus on the best postoperative pain management regimen. In the wake of the opioid epidemic, postoperative pain management is heavily scrutinized. The National Institute of Health estimated over 81,000 individuals died following overdose of any opioids in 2022 alone; of these, over 14,000 deaths were linked to prescription opioids. Thus, strategies to minimize postoperative pain should not only improve patient experience but also lessen the need to escalate to opioid usage.

DETAILED DESCRIPTION:
It would be ideal to create an effective and easily reproducible approach to pain prevention and pain management in men undergoing IPP placement. One highly appealing target would be intracavernosal administration, as there would be no ambiguity regarding delivery of agent at the time of surgery. Thus far, no prospective randomized controlled trials have explored the efficacy of intracavernosal administration of local anesthetic for pain management.

ELIGIBILITY:
Inclusion Criteria:

* Any patient undergoing primary three-piece inflatable penile prosthesis (IPP) placement at Lexington Medical Center

Exclusion Criteria:

* Patients undergoing revision and/or secondary IPP placement
* Patients taking prescribed narcotic medications at the time of IPP surgery
* Patients undergoing concomitant Peyronie's Disease surgery (modeling, plication, grafting) at the time of IPP surgery
* Patients with liver and/or renal disease

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) Scores | Hour 1
  VAS scores range from 0 to 100, with 0 representing no pain or the least desirable state and 100 representing the worst possible pain or the most desirable state. The "score" is the distance in millimeters from the "no pain" end of the 100mm line to the point where the person marks their pain level. Lower scores (0-4mm) indicate no pain, while higher scores (75-100mm) indicate severe pain.
Visual Analogue Scale (VAS) Scores | Hour 4
  VAS scores range from 0 to 100, with 0 representing no pain or the least desirable state and 100 representing the worst possible pain or the most desirable state. The "score" is the distance in millimeters from the "no pain" end of the 100mm line to the point where the person marks their pain level. Lower scores (0-4mm) indicate no pain, while higher scores (75-100mm) indicate severe pain.
Visual Analogue Scale (VAS) Scores | Hour 24
  VAS scores range from 0 to 100, with 0 representing no pain or the least desirable state and 100 representing the worst possible pain or the most desirable state. The "score" is the distance in millimeters from the "no pain" end of the 100mm line to the point where the person marks their pain level. Lower scores (0-4mm) indicate no pain, while higher scores (75-100mm) indicate severe pain.

SECONDARY OUTCOMES:
Cumulative Morphine milligram equivalents (MME) | Day 2
  Cumulative morphine milligram equivalent (MME) is a metric used by healthcare providers to standardize the total potency of all opioid medications a patient is taking. By converting each opioid into a standard value based on morphine, providers can assess a patient's overall risk for overdose and other complications. Higher cumulative MME levels are associated with a greater risk of overdose. For example, doses of 50 MME or more per day increase overdose risk and warrant closer monitoring, while doses of 90 MME or more are considered very high.
Number of calls, messages, or visits to clinic | Day 30
  Physician access line calls, messages to clinic, visits to clinic for postoperative pain within 30 days after surgery
Number of Complications | Day 30
  Complications from intracavernosal injections
Number of Other Complications | Day 30
  Other complications after IPP surgery using the Clavien-Dindo grading scale - The Clavien-Dindo scale is a grading system that categorizes surgical complications based on the treatment required to manage them, providing a uniform and objective way to assess and report post-operative events. It consists of five grades, with Grade I being minor deviations not requiring intervention and Grade V indicating patient death
Serum bupivacaine levels | Hours 1 and 24
  Serum bupivacaine levels at 1 hour and 1 day after surgery - Serum bupivacaine levels are a measurement of the drug in the blood, and the "normal" or safe level varies significantly by the patient's condition, the administration site, and the dose - A 1-mL serum or plasma sample is typically collected in a red-top or green-top tube
Amount of tramadol usage | Hour 24
  Use the lowest dose possible for the shortest time needed. Take your prescribed dose as indicated by your healthcare provider. The maximum dosage is 1 or 2 tablets every 4 to 6 hours, as needed for pain relief.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Terlecki, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the Individual participant data collected during the trial, after deidentification
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Immediately following publication - no end date
Access Criteria: anyone who wishes to access the data